CLINICAL TRIAL: NCT04886661
Title: Correlation of Cervical Lordosis Detected on Cervical X-Ray Images With Clinical, Demographic and MRI Findings
Brief Title: Correlation of Cervical Lordosis Degree Detected on Cervical X-Ray Image With Clinical, Demographic and MRI Findings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Professor, M.D., Haydarpasa Numune Training and Research Hospital
Other Study IDs: HNEAH-KAEK 2021/22
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Neck Pain; Cervical Lordosis; Disk, Herniated
Keywords: neck pain; cervical sagittal balance; trigger points; flex head posture
MeSH Terms: conditions — Neck Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS WITH CHRONIC NECK PAIN: Patients between the ages of 18-65 who are eligible for the inclusion criteria will be included in the study who have cervical X-RAY and cervical MRIs taken in the last 3 months.
  Interventions: Other: CHRONIC NECK PAIN

INTERVENTIONS:
Other: CHRONIC NECK PAIN — Demographic information will be collected. Neck Disability Index will be filled. Physical examination will be performed.

SUMMARY:
In this study we are investigating whether there is a relationship between the lordosis angle measured on cervical X-RAY images on the severity and level of cervical disc herniation detected by cervical MRI, demographic characteristics and the duration and posture of the person's daily life activities.

DETAILED DESCRIPTION:
At least 125 patients between the ages of 18-65 who meet the inclusion criteria with cervical cervical X-RAY and cervical MRIs taken in the last 3 months will be included in the study.

The demographic characteristics of the patients such as age, gender, BMI, job, education level, marital status, as well as the time they spend on head flexion posture, and their screen time will be questioned. The presence of active trigger points in the cervical muscles will be determined by examination (levator scapula, trapeze, longus colli, splenius capitis).

Neck Disability Index will be filled in order to evaluate activities of daily life. Symptom duration and pain level will be evaluated by VAS.

Tangent and Cobb angles will be measured on cervical X-RAY images. Presence of effective lordosis will be recorded.

In cervical MR, disc herniation level, number, degree (bulging, protrusion, extruded disc) its level will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Axial neck pain and / or upper extremity radicular symptoms
* Existing MR and X-Ray radiographs taken within the last 3 months for cervical disc pathologies

Exclusion Criteria:

* A history of trauma,
* Patients with rheumatoid / autoimmune diseases such as rheumatoid arthritis or ankylosing spondylitis,
* A history of Cervical fracture or cervical spine surgery
* History of cancer history, neurological disease
* Muscle weakness
* Presence of Scoliosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 125 Patients with chronic neck pain aged between 18-65 who have their Cervical X-RAY and MRIs being taken within the last 3 months in regards to the inclusion and exclusion criterias.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
C2-C7 COBB ANGLE | 1 week
  MEASURING C2-C7 COBB ANGLE ON LATERAL CERVICAL X-RAY IMAGE
C2-C7 POSTERIOR TANJANT ANGLE | 1 week
  MEASURING C2-C7 POSTERIOR TANJANT ANGLE ON LATERAL CERVICAL X-RAY IMAGE
C2-C7 CERVICAL VERTEBRAL ALIGNMENT (CVA) | 1 week
  C2-C7 CERVICAL VERTEBRAL ALIGNMENT ON LATERAL CERVIKAL X-RAY IMAGE
CERVICAL HERNIATION LEVEL | 1 week
  CERVICAL HERNIATION LEVEL ON CERVICAL MRI
CERVICAL HERNIATION DEGREE | 1 week
  CERVICAL HERNIATION DEGREE ON CERVICAL MRI: BULGING,PROTRUSION, SECESTRATION, EXTRUDATION

SECONDARY OUTCOMES:
DEMOGRAPHIC FINDINGS | 1 week
  AGE
SCREEN TIME | 1 week
  AVARAGE TIME SPENT ON TV, COMPUTER AND MOBILE PHONE DURING A DAY IN HOURS
VISUAL ANALOG SCALE (VAS) | 1 week
  VISUAL ANALOG SCALE SCORE FOR THE NECK PAIN FROM 1-10
NECK DISABILITY INDEX (NDI) | 1 week
  NECK DISABILITY INDEX SCORE
DURATION OF THE NECK PAIN | 1 week
  HOW LONG DOES THE PATIENT FEELS THE NECK PAIN IN MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided